CLINICAL TRIAL: NCT03621631
Title: Real Time Biofeedback Tai Chi Training for Knee Osteoarthritis: A Feasibility Study
Brief Title: Effect of Tai Chi Exercise on Mechanical Joint Loading in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-050; 1K23AT009568-01A1 (NIH)
Record Dates: First submitted 2018-07-31; First posted 2018-08-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; Tai Chi; Biofeedback; External Knee Adduction Moment
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- optimized Tai Chi intervention (Experimental): optimized Tai Chi intervention
  Interventions: Behavioral: Optimized Tai Chi intervention
- traditional Tai Chi intervention (Active Comparator): traditional Tai Chi intervention
  Interventions: Behavioral: Traditional Tai Chi intervention

INTERVENTIONS:
Behavioral: Optimized Tai Chi intervention — Optimized Tai Chi intervention
  Other Names: OTC
  Arms: optimized Tai Chi intervention
Behavioral: Traditional Tai Chi intervention — Traditional Tai Chi intervention
  Other Names: TTC
  Arms: traditional Tai Chi intervention

SUMMARY:
This project is designed to identify the biomechanical mechanisms of Tai Chi (TC) exercise and test a novel optimized TC intervention by modifying newly identified mechanisms for those with knee osteoarthritis (OA) and to assess the changes in mechanical load with the intervention. It combines unique real time torque biofeedback approach, and uses external knee adduction moment (EKAM) as modulation target tailored to TC intervention in this population. The potential benefit from this project is to provide biomechanical insights of TC and this novel TC approach may produce meaningful changes of mechanical load in these patients who can learn and practice safely during this intervention.

DETAILED DESCRIPTION:
Disabilities that arise from typical impairments of knee osteoarthritis (OA) include decreased muscle strength, reduced range of motion, and decreased aerobic cardiovascular function. A large number of individuals with knee OA experience disability and require rehabilitation. Traditional TC intervention has been a promising therapeutic intervention in knee OA, but the efficacy of TC as a knee OA intervention has proven inconclusive presumably because individuals with knee OA perform different TC components (steps) with widely varying mechanical knee joint loads. This variation could be a confounding factor in the way in which TC affects knee OA. Therefore, a feasibility study is proposed here to quantify external knee adduction moment (EKAM) response to the different TC steps, and then determine if it is feasible to use biofeedback of torque acting on the knee to modify some TC steps so as to reduce the EKAM they produce. Those TC steps whose EKAM can be easily reduced below mean EKAM during walking and those already below that level will constitute an optimized form of TC for knee OA; the remainder will be discarded. A phase 1 randomized controlled trial will be conducted to compare the optimized TC intervention to traditional TC training in reducing EKAM. The proposed research represents the first study to identify the biomechanical mechanisms of TC and to target EKAM by using a real-time biofeedback approach to manipulate EKAM during TC performance.

ELIGIBILITY:
Inclusion Criteria:

* OA participants will be diagnosed based on the American College of Rheumatology classification criteria.
* Knee pain average level > 3 cm on a 10 cm visual analog scale,
* Kellgren / Lawrence scale of 2-3 on radiographs.
* Pain/tenderness over the medial region or lateral region of the knee on physical examination.
* The participants will have 40 years of age or older and have no TCC experience prior this study.

Exclusion Criteria:

* a history of lower extremity joint replacement
* intra-articular knee injection (steroid, hyaluronic acid) within the previous 6 months
* systemic rheumatoid arthritic condition affecting the knee clinically or radiographically,
* report of any of the following health problems (heart condition, chest pain during periods of activity or rest)
* currently seeking or receiving physical therapy for knee OA,
* having a medical condition precluding the participant from undergoing physical activity or biomechanical gait analysis.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
change from baseline knee joint mechanical load at 4 weeks | baseline and 4 weeks
  knee joint mechanical load will be measured by using high speed cameras and force plates to estimate external knee adduction moment (EKAM)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Health San Antonio, Rehabilitation Biomechanics Lab, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary outcome measure will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 6 month of study completion
Access Criteria: Data access requests will be reviewed by an external independent review panel.

REFERENCES:
- [Derived] Yang F, Markides K, Reistetter TA, Moore AA, Liu W. Effects of Optimal Tai Chi forms in alleviating knee pain among Hispanic people with knee osteoarthritis: A case series. Complement Ther Clin Pract. 2025 May;59:101961. doi: 10.1016/j.ctcp.2025.101961. Epub 2025 Feb 12. PMID 39961273